CLINICAL TRIAL: NCT04814953
Title: HRQoL and Development of Health Utilities in Patients With Keratinocyte Carcinomas
Brief Title: HRQoL Keratinocyte Carcinomas
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BC-5344
Record Dates: First submitted 2020-06-16; First posted 2021-03-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma; Actinic Keratoses
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Keratosis, Actinic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Basal cell carinoma patients: Patients with basal cell carcinoma in history (up to 10 years before inclusion) with or without squamous cell carcinoma or actinic keratosis but no other skin cancers (melanoma or non-melanoma skin cancer)
  Interventions: Other: questionnaires
- Squamous cell carcinoma patients: Patients with squamous cell carcinoma in history (up to 10 years before inclusion) with or without basal cell carcinoma or actinic keratosis but no other skin cancers (melanoma or non-melanoma skin cancer)
  Interventions: Other: questionnaires
- Patients with actinic keratoses: Patients with actinic keratosis in history (up to 10 years before inclusion) with or without basal cell carcinoma or squamous cell carcinomas but no other skin cancers (melanoma or non-melanoma skin cancer)
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — EQ-5D-5L questionnaire questioning their overall health on five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). In addition patients will have to fill in the generic 15D questioning 15 specific dimensions on 5 levels as well as the BaSQoL, which is a disease specific questionnaire for patients with KC. The Time-trade off task is the final question.

SUMMARY:
Rationale: Keratinocyte skin cancer is known to influence the HRQoL in a specific way. Derived utility values are required for cost-effectiveness analyses of new interventions. However there is no sensitive tool to capture HRQoL that translates into utilities available.

Objective: To document the exact HRQoL in patients with in KC using the generic EQ-5D-5L questionnaire, as well as the TTO, 15D and the BaSQoL questionnaire, and to develop health utilities based on these tools.

Study design: Longitudinal observational study (at time 0 and time 0 +12 months).

Study population: Patients aged ≥18 years consulting a dermatologist or their GP for diagnosis, treatment or follow-up of a (pre)malignant skin lesion(s).

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion criteria

1. Patients with one or more premalignant lesion or KC diagnosed by a dermatologist or by histopathology untill 10 years previous to inclusion.

Exclusion criteria

1. Patient is younger than 18 years old or unable to provide consent.
2. Patient is unable to remember the diagnosis or symptoms of their KC or premalignant lesion upon request by the doctor.
3. Patient was diagnosed with a melanoma or another NMSC.
4. Patient is unable to understand the task and questionnaires.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Department of Dermatology of the University Hospital of Ghent and the Erasmus MC Rotterdam. In addition, patients in other hospitals and dermatology clinics will be asked to participate. Two general practitioners will also include patients with a KC or actinic keratoses.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health utility (by using a time trade off questionnaire) | 1 year
  Utilities as determined by the time trade off, this is a technique used to measure the quality of life that a person or group is experiencing. An individual will be presented with a set of directions such as, and the result will be a health utility index between 0-1. Lower scores mean less HrQoL.
Health utility (by using the 15D questionnaire) | 1 year
  Utilities as determined by the 15D questionnaire, a generic questionnaire developed to determine a health utility index between 0-1. Lower scores mean less HrQoL.
Health utility (by using the EQ-5D-5L questionnaire) | 1 year
  Utilities as determined by the EQ-5D questionnaire, a generic questionnaire developed to determine a health utility index between 0-1. Lower scores mean less HrQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Hoorens, MD, PhD, Principal Investigator — Ghent University Hospital, Department of Dermatology
Locations (2):
- Department of Dermatology, Ghent University Hospital, Ghent, Belgium
- MC Rotterdam Department of Dermatology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No